CLINICAL TRIAL: NCT05249374
Title: A Randomized, Double-blind, Active Drug-controlled, Dose-escalation Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of r-HSA in Patients With Cirrhosis and Ascites
Brief Title: Recombinant Human Serum Albumin in Patients With Liver Cirrhosis and Ascites Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protgen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rHSA 2020-2
Record Dates: First submitted 2022-01-27; First posted 2022-02-21 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Hepatic Ascites
MeSH Terms: interventions — recombinant human serum albumin-heme; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 10 g/ bottle (20%, 50 mL)
  Interventions: Drug: Recombinant Human Serum Albumin
- test group (Experimental): 10 g/bottle (20%, 50 mL)
  Interventions: Drug: Human serum albumin

INTERVENTIONS:
Drug: Recombinant Human Serum Albumin — 10 g/bottle (20%, 50 mL)
  Arms: Control group
Drug: Human serum albumin — 10 g/bottle (20%, 50 mL)
  Arms: test group

SUMMARY:
This trial adopts a randomized, double-blind, positive drug-controlled, dose-escalated phase Ib clinical study evaluating the safety, tolerability, pharmacokinetic characteristics and preliminary effectiveness of recombinant human serum albumin in patients with liver cirrhosis and ascites

subjects (both male and female) were screened and enrolled to the three dose levels of 10g, 20 g,and 30 g according to the principle of dose escalation, and 8 out of 12 subjects in each dose group One patient received the test drug, and 4 received a positive drug.

DETAILED DESCRIPTION:
In this Phase Ib clinical trial, randomized, double-blind, positive-controlled, dose-increasing design was employed to enroll cirrhosis ascites patients and evaluate safety, tolerability, PK characteristics, PD characteristics and preliminary efficacy at different dose levels of recombinant human serum albumin.

Three dose groups (10 g/day, 20 g/day, 30 g/day) were set up in this study, and they were escalated from the lowest to the highest dosage. It is planned to enroll 12 subjects in each dose group, with 8 of 12 subjects in each dose group receiving the investigational product and 4 of 12 subjects receiving the comparator product intravenously once a day for 14 days or up to serum albumin ≥ 35 g/L ( whichever occurs first ), to investigate the safety, tolerability, immunogenicity, PK characteristics, PD characteristics and preliminary efficacy in repeated usage of recombinant human serum albumin.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the experimental treatment plan and visit plan, voluntarily enroll in the group, and sign the informed consent in person;
2. Age ≥18 years old and <65 years old on the day of signing the informed consent, no gender limitation; Body mass index (BMI) ranged from 18.0 kg/m2 to 29.0 kg/m2 (including boundary values);
3. Patients clinically diagnosed as decompensated cirrhotic ascites with ascites grade 1-2 and serum albumin (ALB) <30 g/L confirmed by abdominal ultrasonography during screening period;
4. Men and women of child-bearing age with fertility (childbearing age women including premenopausal women and 2 years after menopause women) from willing to sign a consent form began to experiment with drugs within 3 months after the last delivery effective precautions (take a condom, contraceptive sponge, contraceptive gel, diaphragm, intrauterine device, oral or injectable contraceptives, subcutaneous preparetions Agent, etc.); Women of reproductive age must have a negative pregnancy test no later than 7 days before the first investigational drug is administered.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for inclusion:

1. Patients with malignant ascites;
2. People who have a known history of allergy/allergic reaction to yeast or yeast-derived products or are allergic to any component of the study product; Patients with an allergic constitution (multiple drug or food allergy), a history of allergic to biological products, or a history of severe systemic allergic reaction caused by other reasons, and the investigator judges that they are not suitable for treatment with experimental drugs;
3. The patient has the following abnormal laboratory tests:

   Bone marrow function: absolute value of neutrophils (ANC) <1.0×109/L (1000/mm3); Platelet (PLT) <20×109/L (2×104/mm3); Hemoglobin (HGB) <7.0 g/dL;Liver function: alanine aminotransferase (ALT) > 5×ULN (upper normal value); Aspartate aminotransferase (AST) > 5×ULN; Serum bilirubin (T-Bil) >3× upper normal value (ULN);Renal function: serum creatinine >2× upper normal value (ULN); Positive urine protein and ineligible to participate in the test judged by the investigator; coagulation function: prothrombin activity <40%;
4. Active cardiovascular disease or history at the time of screening, or other conditions that the investigator determined were not suitable for human serum albumin therapy, including but not limited to hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg), Researchers determine drug control is good and stable condition except), severe anemia, heart disease, acute severe lung or structural heart disease, severe arrhythmia, normal blood volume (or high blood volume) of decompensated heart failure, unstable angina, nearly six months prior to screening the myocardial infarction, require drug treatment of tachycardia/slow, three degree atrioventricular block, etc.;
5. At the time of screening, there was a history of active metabolic system disease or other renal injury that the investigator determined was unsuitable for serum albumin treatment, including but not limited to renal/postrenal anuria, hepatorenal syndrome (HRS), chronic kidney disease, hepatitis B related nephropathy, etc.;
6. Patients with the following active concurrent diseases during screening, including but not limited to, Pulmonary edema, bleeding tendency, or active bleeding disease, sustained or active infection (including active spontaneous bacterial peritonitis (SBP)), according to West - Haven classification standard diagnosis of hepatic encephalopathy grade III or IV level, portal venous tumor emboli/blood clots, circulation dysfunction after abdominal puncture, ultrasound and other imaging examination of biliary obstructive disease Disease, thyroid dysfunction (grade 3 and above according to NCI CTCAE version 5.0);
7. Patients with previous history of upper gastrointestinal bleeding within 1 month or gastrointestinal bleeding within 3 months (≥2 times) or high risk of bleeding during the study as assessed by the investigator;
8. Patients with active malignancies (including hepatocellular carcinoma [HCC]) at the time of screening, or with a history of malignant tumors within 5 years (except cancer in situ, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ and other very low-risk malignancies of cervical or breast cancer undergoing curative treatment);
9. Those who have received corticosteroids or human plasma preparations (including human serum albumin preparations) within 20 days prior to the first administration of the investigational drug; Those with a history of organ transplantation; Those requiring or planning to undergo invasive tests or treatment during the study period;
10. Participating in or participating in clinical trials of other new drugs or medical devices and using investigational drugs/investigational treatments within 30 days prior to screening; Prior participation in clinical trials of recombinant human serum albumin;
11. HIV antibody test positive, or syphilis (defined as positive syphilis antibody test and positive retin test);
12. Pregnant or lactating women;
13. Other reasons that the researcher considers inappropriate to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
TEAE | 57 days
  Adverse events will be coded using MedDRA (International Dictionary of Medical Terms)., TEAEs related to test drugs were summarized and analyzed according to SOC and PT, and the number of occurrences and the incidence were calculated.
SAE | 57 days
  Adverse events will be coded using MedDRA (International Dictionary of Medical Terms). SAEs related to test drugs were summarized and analyzed according to SOC and PT, and the number of occurrences and the incidence were calculated.

SECONDARY OUTCOMES:
AUC0-last | 57 days
  Within 1 hour before administration of D1, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes);
  If subject has completed 14 days of treatment, then:
  Within 1 hour before administration of D2~D13, immediately after administration (+1 min); D14: within 1 hour before administration, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes); D15, D16, D17, D29 (±3 days), D57 (±5 days).
  If the 14-day treatment has not been completed, then:
  Before drug withdrawal: receive 2 PK blood sample collections within 1 hour before administration and immediately after administration (+1 min) each day; After drug withdrawal: from the day of drug withdrawal, collect PK blood samples once for 3 consecutive days.
Pharmacokinetic characteristics | 57 day
  Within 1 hour before administration of D1, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes);
  If subject has completed 14 days of treatment, then:
  Within 1 hour before administration of D2~D13, immediately after administration (+1 min); D14: within 1 hour before administration, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes); D15, D16, D17, D29 (±3 days), D57 (±5 days).
  If the 14-day treatment has not been completed, then:
  Before drug withdrawal: receive 2 PK blood sample collections within 1 hour before administration and immediately after administration (+1 min) each day; After drug withdrawal: from the day of drug withdrawal, collect PK blood samples once for 3 consecutive days.
Albumin concentration of D15 | 1 day
  Collect blood samples on the fifteenth day and determine the albumin concentration on the fifteenth day.
Albumin concentration of D29 | 1 day
  Collect blood samples on the 29th day(±3 days) and determine the albumin concentration on the 29th day.
Albumin concentration of D57 | 1 day
  Collect blood samples on the 57th day（±5 days） and determine the albumin concentration on the 57th day.
t1/2 | 57 days
  Within 1 hour before administration of D1, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes);
  If subject has completed 14 days of treatment, then:
  Within 1 hour before administration of D2~D13, immediately after administration (+1 min); D14: within 1 hour before administration, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes); D15, D16, D17, D29 (±3 days), D57 (±5 days).
  If the 14-day treatment has not been completed, then:
  Before drug withdrawal: receive 2 PK blood sample collections within 1 hour before administration and immediately after administration (+1 min) each day; After drug withdrawal: from the day of drug withdrawal, collect PK blood samples once for 3 consecutive days.
CL | 57 days
  Within 1 hour before administration of D1, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes);
  If subject has completed 14 days of treatment, then:
  Within 1 hour before administration of D2~D13, immediately after administration (+1 min); D14: within 1 hour before administration, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes); D15, D16, D17, D29 (±3 days), D57 (±5 days).
  If the 14-day treatment has not been completed, then:
  Before drug withdrawal: receive 2 PK blood sample collections within 1 hour before administration and immediately after administration (+1 min) each day; After drug withdrawal: from the day of drug withdrawal, collect PK blood samples once for 3 consecutive days.
Cpost-Cpre | 14 days
  Calculate the ratio of serum albumin concentration to C0 at each time point, and calculate the difference of albumin concentration before and after each intravenous administration
Plasma colloid osmotic pressure | 17 days
  D1 within 1 hour before administration, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes);
  If the 14-day treatment cycle is completed, then:
  Within 1 hour before administration of D2~D13, immediately after administration (+1 min); D14: within 1 hour before administration, immediately after administration (+1 min), 2 hours (±5 minutes), 10 hours (±30 minutes); D15, D16, D17.
  If discontinuation of 14-day treatment cycle is not completed, then:
  Before drug withdrawal: 2 blood samples were collected within 1 hour before each administration and immediately after the administration (+1 min); After drug withdrawal: From the day of drug withdrawal, collect PD blood samples once for 3 consecutive days.
the Anti-Drug antibody (ADA) of rHSA | 57 days
  All subjects in this trial who received at least 1 intravenous dose, regardless of when they ended treatment, were required to visit D1 before intravenous administration of the investigational drug, D8, D15, D29, D57, and at the early withdrawal visit (if any). ADA blood samples were collected, and the sample collection time window was the same as the time window of the current visit. Immunogenicity was assessed by assessing the incidence and titers of anti-rHSA, if applicable.
the Anti-Drug antibody (ADA) of HCP | 57 days
  All subjects in this trial who received at least 1 intravenous dose, regardless of when they ended treatment, were required to visit D1 before intravenous administration of the investigational drug, D8, D15, D29, D57, and at the early withdrawal visit (if any). ADA blood samples were collected, and the sample collection time window was the same as the time window of the current visit. Immunogenicity was assessed by assessing the incidence and titers of anti-host protein (HCP) ADAs, if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Chen, Ph.D, Study Director — Peking Union Medical College Hospital
Locations (1):
- Shenzheng Protgen Ltd, Guangdong, Shenzheng, China

IPD SHARING:
Plan to Share IPD: No